CLINICAL TRIAL: NCT05086601
Title: A Cohort of Molecular Characteristics and Prognosis of Colorectal Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Sponsor
Other Study IDs: CRCC2021
Record Dates: First submitted 2021-09-23; First posted 2021-10-21 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-03

CONDITIONS: Colorectal Cancer; Surgery
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — The specimens include primary tumor tissue, adjacent tissues, normal mucosa tissue, and peripheral venous blood. Tissue samples will be used for multiple omics tests, including genome, transcriptome, proteome, etc. Blood samples are used for tumor markers, immunology and other tests.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: colorectal cancer surgery — Any surgery for primary tumor of colorectal cancer, including palliative resection, simple bowel stoma and exploratory surgery.

SUMMARY:
This study aims to establish a colorectal cancer cohort, collect clinicopathological information, collect biological samples for multi-omics testing, and perform relevant analysis, to predict the prognosis of colorectal cancer, guide the diagnosis and treatment of colorectal cancer and the formulation of health policies.

DETAILED DESCRIPTION:
In this study, the investigators will establish a database to collect clinical pathological information, based on the medical data system of participating medical centers. The investigators will also collect corresponding tumor specimens and perform multiple omics tests such as genome, transcriptome, and proteome. The investigators will aggregate these data into a special database, and use appropriate methods to conduct big data analysis, to predict prognosis, guide diagnosis and treatment, and assist in formulating health policies.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically diagnosed as colorectal cancer
* Receiving any surgery of primary tumor, including palliative resection, simple enterostomy and exploratory surgery

Exclusion Criteria:

* The patient refused to join the study
* The patient refused to collect the biological sample
* The patient refused to follow up

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients pathologically diagnosed as colorectal cancer, and receiving any surgery of primary tumor, including palliative resection, simple enterostomy and exploratory surgery
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-09-09 (Estimated); Study Completion 2022-09-09 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival time | 2 yeas after surgery
  For patients received radical resection of colorectal cancer, disease-free survival time is defined as time from the surgery to any recurrence of disease or death, recorded in months.

SECONDARY OUTCOMES:
Overall survival time | 2 yeas after surgery
  Overall survival time is defined as time from the surgery to death, recorded in months.
Pathological TNM stage | 1 month after surgery
  The pathological TNM stage included the pathological T stage, pathological N stage and M stage. The pathological T and N stage is decided according to the removed specimen of the primary tumor by the pathologist after surgery. The M stage is decided according to the imaging tests as CT, MRI and PET-CT.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No